CLINICAL TRIAL: NCT01254981
Title: Randomized Clinical Comparative Study of the Nobori and the Cypher Stents in Unselected Subjects With Ischemic Heart Disease
Brief Title: SORT-OUT V - Randomised Clinical Comparative Study of the Nobori and the Cypher Stent.
Acronym: SORT-OUT V
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Terumo Europe N.V. (Industry); Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Evald Hoej Christiansen, MD. DMSc, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M-20090103
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Coronary Artery Disease; Angina Pectoris
Keywords: Percutaneous coronary intervention; DES; Angina pectoris; Stent
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nobori (Experimental): Percutaneous coronary intervention with implantation of coronary stent (Nobori)
  Interventions: Procedure: Percutaneous coronary intervention (PCI)
- Cypher (Experimental): Percutaneous coronary intervention with implantation of coronary stent (Cypher)
  Interventions: Procedure: Percutaneous coronary intervention (PCI)

INTERVENTIONS:
Procedure: Percutaneous coronary intervention (PCI) — Implantation of coronary stent
  Other Names: PCI; PTCA

SUMMARY:
To perform a randomized comparison between the Cypher Select+ stent and the Nobori stent in the treatment of unselected patients with ischaemic heart disease.

DETAILED DESCRIPTION:
All patients to be treated with one or several drug-eluting coronary stents at one of the four heart centers in Odense, Skejby, Aalborg and Varde can be included in the study. All patients enrolled in the study will be hospitalized at one of the heart centers mentioned. Patients will not be recruited via advertisements.

The study is designed as a non-inferiority study, where the objective is to prove that Nobori is Δ0 poorer as a maximum than Cypher select+. The nine-month event rate (cardiac death, MI and/or TVR) in the Cypher stent group of SORT OUT 3 was 3.0%

The calculation of power below has been made under the following assumptions:

P (Cypher) = 0.03

There is no good estimate for the event rate related to the Nobori stent. α = 0.05 - one-sided

1-β = 0.80

Based on the various values of Δ0 the necessary number of patients, N, in each group can be calculated (StudySize Version 2.0.4, Creostat):

* Δ0 *N in each group
* 0.0025 *57,589
* 0.005 *14,397
* 0.010 *3,599
* 0.015 *1,599
* 0.020 *900

According to the above assumptions, a total of 900 patients must be included in each group in order to reject a null hypothesis that the event rate in the Nobori group is more than 2 percentage points (0.02) poorer than the event rate in the Cypher group or that Nobori is inferior to Cypher, (H0: pNobori - pCypher ≥ Δ0 = 0.02). The alternative hypothesis (HA: pN - pS < Δ0) provides that Nobori is non-inferior to Cypher - with the selected limit for non-inferiority.

Assuming an inclusion rate of 200 patients per month, it will be possible to include 2000 patients in 10 months.

Power is almost 0.9 if the inclusion is increased to a little over 2400.

Organization

The study is headed by a steering committee, in which PCI operators will participate from each of the participating sites.

Evald Høj Christiansen, Aarhus, will be Principal Investigator. At present, the other members of the steering committee are: Jens Flensted Lassen (chairman), Leif Thuesen, Jan Ravkilde, Hans-Henrik Tilsted, Per Thayssen and Lisette Okkels Jensen. All members of the steering committee will be given full access to the database and will take part in the interpretation of data.

The study secretariat and the randomization computer are localized at the Department of Cardiology, [Hjertemedicinsk Afdeling], Aarhus University Hospital, Skejby.

ELIGIBILITY:
Inclusion Criteria:

All patients eligible for treatment with one or several drug-eluting coronary stents at one of the four heart centers in Odense, Skejby, Aalborg or Varde can be included in the study.

The patients will be treated in accordance with the criteria applicable at the individual sites. The indication for using DES varies slightly between the four sites, as the indication for implantation of DES is based on clinical and angiographic criteria with the financial constraints applying at the individual site. Basically, DES will be chosen instead of BMS in patients with an estimated increased risk of restenosis, in patients with the following stenosis types: Long lesions, lesions in small vessels, bifurcations, ostial lesions, in-stent restenoses and stenosis in the proximal segment of the anterior descending branch. Furthermore, DES will also be chosen for diabetics and in the left main.

Exclusion Criteria:

* The patient does not wish to participate
* The patient is participating in other randomized stent studies
* Life expectancy < 1 year
* Allergic to Aspirin, clopidogrel, prasugrel or ticlopidin
* Allergic to sirolimus or biolimus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2504 (Actual)
Dates: Start 2009-07; Primary Completion 2011-01 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Primary outcome | Within 9 months
  Major Adverse Cardiac Events, such as cardiac death, myocardial infarction, stent thrombosis or target lesion revascularisation: repeated revascularisation of an index lesion at PCI or bypass surgery

SECONDARY OUTCOMES:
Secondary outcome
  * Device success rate defined as the frequency of a successful implantation of the study stent in all the stenoses scheduled to be treated with residual stenosis < 20
  * Procedural success rate defined as the frequency of successful implantation of the study stent in all the stenoses scheduled to be treated with residual stenosis < 20% and without serious complications (MACE = Major Adverse Coronary Events))
  * Procedural time defined as time from guiding catheter in to guiding catheter out
  * X-ray time
  * Use of contrast medium
Major Adverse Coronary Events | 30 days
  Cardiac death, myocardial infarction, target vessel revascularisation: repeated revascularisation of an index lesion at PCI or bypass surgery
Target lesion revascularisation defined as repeated revascularisation of an index lesion at PCI or bypass surgery. | 9 and 12 months and 3 years
Death | 30 days and 9 months
Acute Myocardial Infarction | 30 days and 9 months
Stent thrombosis | 12, 24 and 36 months
  Defined in accordance with the ARC definition of stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Evald H Christiansen, MD, Principal Investigator — Aarhus University Hospital Skejby
Locations (3):
- Denmark (3):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus University Hospital, Skejby, Aarhus N
  - Odense University Hospital, Odense

REFERENCES:
- [Derived] Christiansen EH, Jensen LO, Thayssen P, Tilsted HH, Krusell LR, Hansen KN, Kaltoft A, Maeng M, Kristensen SD, Botker HE, Terkelsen CJ, Villadsen AB, Ravkilde J, Aaroe J, Madsen M, Thuesen L, Lassen JF; Scandinavian Organization for Randomized Trials with Clinical Outcome (SORT OUT) V investigators. Biolimus-eluting biodegradable polymer-coated stent versus durable polymer-coated sirolimus-eluting stent in unselected patients receiving percutaneous coronary intervention (SORT OUT V): a randomised non-inferiority trial. Lancet. 2013 Feb 23;381(9867):661-9. doi: 10.1016/S0140-6736(12)61962-X. Epub 2013 Jan 30. PMID 23374649